CLINICAL TRIAL: NCT02503124
Title: Wake and Bright Light Therapy for Depression Among Admitted Patients
Brief Title: Effect of a Single Nights' Wake Followed by Bright Light Therapy for Severe Depression
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 and re-organisation at the hospital
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Steinn Steingrimsson, MD, PhD, resident in psychiatry, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CB001
Record Dates: First submitted 2015-07-10; First posted 2015-07-20 (Estimated); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chronobiological intervention (Experimental): Single night's wake therapy followed by bright light therapy for a week as add-on treatment to treatment as usual.
  Interventions: Behavioral: Single night's wake therapy; Device: Bright light; Other: Treatment as usual - inpatient care; Drug: Treatment as usual - medicine
- Control (Active Comparator): Treatment as usual including a private educational meeting in sleep hygiene.
  Interventions: Other: Treatment as usual - inpatient care; Other: Informative meeting; Drug: Treatment as usual - medicine

INTERVENTIONS:
Behavioral: Single night's wake therapy — Eligible patients are assisted in maintaining total sleep deprivation during one night
  Other Names: Sleep deprivation
  Arms: Chronobiological intervention
Device: Bright light — Bright light according to patients´ own circadian rhythm each morning for a week.
  Arms: Chronobiological intervention
Other: Treatment as usual - inpatient care — All patients are admitted due to severe depression and are under observation and most receive antidepressive medication and if necessary anxiolytic/antipsychotic medication.
Other: Informative meeting — A short sleep hygiene consultation.
  Arms: Control
Drug: Treatment as usual - medicine — Since all patients are admitted due to a severe mental illness, they will receive medication according to indication. Most patients have already tried more than one antidepressant at the time of admission. In cases of severe anxiety, anxiolytics are prescribed but this is kept to a minimum.

SUMMARY:
A randomized controlled trial comparing wake therapy (single night) followed by bright light therapy to treatment as usual.

ELIGIBILITY:
Inclusion Criteria:

* Depressive episode requiring admission to a psychiatric hospital (including unipolar and bipolar depression).

Exclusion Criteria:

* Psychotic symptoms/agitation
* Compulsory admission
* Confusion
* Active substance use disorder
* Eye disease preventing bright light therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-07; Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
MADRS-S score reduction of 50% | One week
  Montgomery Asberg Depression Rating Scale

SECONDARY OUTCOMES:
MADRS-S score at discharge | Participants will be followed at discharge, an expected average of 2-3 weeks
  Montgomery Asberg Depression Rating Scale
MADRS-S score at follow-up | 10-14 weeks
  Montgomery Asberg Depression Rating Scale
ISI score score at discharge | Participants will be followed at discharge, an expected average of 2-3 weeks
  Insomnia Severity Index - Self administered scale of sleep quality
ISI score score at follow-up | 10-14 weeks
  Insomnia Severity Index - Self administered scale of sleep quality
ISI score reduction of 50% | One week
  Insomnia Severity Index - Self administered scale of sleep quality
Length of stay | The number of days between admission and discharge
  Patients will be followed up 10-14 weeks after discharge and the total number of days in inpatient services calculated.
Re-admission | 10-14 weeks
CGI score | One week
  Clinical global impression
CGI score | 10-14 weeks
  Clinical global impression
Medication use | 10-14 weeks
  The use of antidepressants, anxiolytics or other psychiatric medication will be registered at follow-up. The number of patients using more than one medication and the dosage will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Steinn Steingrimsson, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided